CLINICAL TRIAL: NCT00071786
Title: Family Study of Affective and Anxiety Spectrum Disorders
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030211; 03-M-0211
Record Dates: First submitted 2003-10-30; First posted 2003-10-31 (Estimated); Last update posted 2025-12-31 (Actual); Status verified 2025-11-14

CONDITIONS: Mood Disorders; Sleep Disorders; Migraine
Keywords: Bipolar; Migraine; High Risk Study; Mobile Technologies; Sleep; Natural History
MeSH Terms: conditions — Mood Disorders; Sleep Wake Disorders; Migraine Disorders

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: All study participants fall into one group for this observational family study regardless of diagnosis.

SUMMARY:
This study will examine how depression, anxiety, and migraine run in families. It will help in defining the risk factors for physical, mental, and health problems-as well as define ways that those problems may be prevented and treated.

A broad range of ages among family members will be included to evaluate the patterns of how these disorders are expressed throughout people's lives. Children of all ages will be included, and those ages 8 to 17 will be interviewed directly.

Assessments will be collected through criteria of the Diagnostic and Statistical Manual of Mental Disorders IV as well as the spectrum, or range, of mood disorders and co-existing conditions. A member of the study team will visit the participants at home or will do an interview by telephone. Participation will take approximately 3 to 4 hours. Children will complete questionnaires given by the research team as well as questionnaires that they will do by themselves. The questions will pertain to the children's health, including physical and mental health and medical history, social relationships, problems, skills, and ways of dealing with important or stressful issues in their lives. These questionnaires will take up to 1 hour to complete.

Health history gathered from adult participants will pertain to height, weight, exercise, and general function. Women will be asked about the use of oral contraceptives, estrogen, and progesterone. In addition, there will be questionnaires on personality and temperamental traits, that is, behavior and impulsiveness. Questions will also involve social intuition, family and other environmental factors, general functioning, and basic demographics such as ethnicity, race, socioeconomic status, marital status, education level, and employment history.

Families enrolled in this phase of the research will be invited to participate in the next phase. There would be follow-up to evaluate the development of mood disorders, subtypes, and syndromes across the lifespan.

DETAILED DESCRIPTION:
Objective:

The chief goal of this study is to identify the endophenotypes of the spectrum of mood disorders using the methods of genetic epidemiology, developmental psychopathology and clinical psychiatry/psychology. The major research questions focus on the specificity of familial transmission of the mood disorder spectrum (i.e., symptoms, symptom clusters, subtypes) and the role of comorbidity with anxiety disorders and migraine syndromes in defining subtypes of mood disorders.

Study Population:

We propose to recruit 800 probands with bipolar I, bipolar II, major depression, panic/GAD, phobias, migraine, and unaffected controls, ascertained through both psychiatric and non-psychiatric clinical settings and systematic community samples, in order to enhance generalizability to the population. Approximately 2750 first-degree adult relatives and spouses, 350 child offspring (ages 7-17) will comprise the family study component.

Design:

This study employs a retrospective cohort family study for the association between mood and other mental and physical disorders in probands and their relatives. Probands and relatives will be evaluated using structured diagnostic interviews and standardized diagnostic criteria followed by clinical validation interviews and diagnostic consensus procedures. Assessment instruments will collect information on the DSM-IV criteria as well as the spectrum of mood disorders and comorbid conditions. In addition, DNA will also be collected from participants. A subset of families will also complete electronic diaries and measures of light exposure and activity in this protocol, and will be invited to participate in another protocol to undergo more comprehensive evaluation of clinical, laboratory, and other functional domans to identify biologic markers and endophentypes for mood and related disorders. Data from the two protocols will be linked. A subset of families will also be followed forward over time.

Outcome Measures:

The primary outcome measure is the familial aggregation of mood disorder subtypes and their co-aggregation with migraine and anxiety disorders with diagnoses based on clinical review of the diagnostic interviews, family history information and clinical evaluation of study participants when relevant using traditional family study measures of association. Secondary outcomes include associations between mood disorders with the data collected from laboratory, biological, and functional assessments that have been collected as part of the clinical study and their familial correlations. Moving forward, these data will be collected as part of a new protocol and linked with the interview and mobile assessment data collected in this protocol.

ELIGIBILITY:
* Since this study is based on systematic recruitment from the local community and other non-clinical settings such as screening protocols from volunteers, there are no specific diagnostic inclusion and exclusion criteria. However, the study targets individuals with mood spectrum conditions and migraine. Criteria for the specific subgroups of mood and anxiety disorders are presented in Table 1. Individuals who do not meet criteria are classified as controls.

INCLUSION CRITERIA:

1. the ability to comprehend the interview, and
2. probands must agree to contact at least two relatives (contacting relatives is not required in cases where the participant is enrolled in just the mobile technologies assessments (EMA and Actigraphy).

   EXCLUSION CRITERIA:

   The only exclusion criteria include impaired ability to comprehend the interview or inability to read.

   SPECIFIC INCLUSION AND EXCLUSION CRITERIA BY PROBAND GROUP:

   GENERAL INCLUSION CRITERIA:

   The only inclusion criteria for the study are that the person be English-speaking and ability to read and comprehend the interview.

   BIPOLAR I INCLUSION CRITERIA:

   Lifetime history of DSM-IV Bipolar I or Manic Episode

   BIPOLAR II INCLUSION CRITERIA:

   Lifetime history of DSM-IV Bipolar II with duration of hypomania reduced to 2 or more days (according to RDC)

   MAJOR DEPRESSION INCLUSION CRITERIA:

   Lifetime history of at least 2 episodes of DSM-IV Major Depression

   PANIC/GAD INCLUSION CRITERIA:

   Lifetime history of DSM-IV diagnosis for Panic Disorder or GAD

   PHOBIAS INCLUSION CRITERIA:

   Lifetime history of DSM-IV diagnosis for social anxiety disorder, agoraphobia, or specific phobias (greater than or equal to 3)

   MIGRAINE INCLUSION CRITERIA:

   Lifetime history of IHS migraine with or without Aura

   GENERAL EXCLUSION CRITERIA:

   The only exclusion criteria include impaired ability to comprehend the interview or inability to read.

Ages: 7 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Community Sample
Sampling Method: Non-Probability Sample
Enrollment: 1944 (Actual)
Dates: Start 2004-05-21 (Actual)

PRIMARY OUTCOMES:
diagnostic interviews, family history information and clinical evaluation of study participants | Lifetime
  Diagnoses, Symptoms, Impairment, Biologic parameters

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen R Merikangas, Ph.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kendell RE. Clinical validity. Psychol Med. 1989 Feb;19(1):45-55. doi: 10.1017/s0033291700011016. PMID 2657832
- [Background] Tsuang MT, Faraone SV, Lyons MJ. Identification of the phenotype in psychiatric genetics. Eur Arch Psychiatry Clin Neurosci. 1993;243(3-4):131-42. doi: 10.1007/BF02190719. PMID 8117756
- [Background] Smoller JW, Tsuang MT. Panic and phobic anxiety: defining phenotypes for genetic studies. Am J Psychiatry. 1998 Sep;155(9):1152-62. doi: 10.1176/ajp.155.9.1152. PMID 9734536
- [Derived] Stapp EK, Zipunnikov V, Leroux A, Cui L, Husky MM, Dey D, Merikangas KR. Specificity of affective dynamics of bipolar and major depressive disorder. Brain Behav. 2023 Sep;13(9):e3134. doi: 10.1002/brb3.3134. Epub 2023 Aug 13. PMID 37574463
- [Derived] Glaus J, Cui L, Hommer R, Merikangas KR. Association between mood disorders and BMI/overweight using a family study approach. J Affect Disord. 2019 Apr 1;248:131-138. doi: 10.1016/j.jad.2019.01.011. Epub 2019 Jan 15. PMID 30731280
- [Derived] Lamers F, Swendsen J, Cui L, Husky M, Johns J, Zipunnikov V, Merikangas KR. Mood reactivity and affective dynamics in mood and anxiety disorders. J Abnorm Psychol. 2018 Oct;127(7):659-669. doi: 10.1037/abn0000378. PMID 30335438
- [Derived] Glaus J, Van Meter A, Cui L, Marangoni C, Merikangas KR. Factorial structure and familial aggregation of the Hypomania Checklist-32 (HCL-32): Results of the NIMH Family Study of Affective Spectrum Disorders. Compr Psychiatry. 2018 Jul;84:7-14. doi: 10.1016/j.comppsych.2018.03.010. Epub 2018 Apr 3. PMID 29655654
- [Derived] Lamers F, Cui L, Hickie IB, Roca C, Machado-Vieira R, Zarate CA Jr, Merikangas KR. Familial aggregation and heritability of the melancholic and atypical subtypes of depression. J Affect Disord. 2016 Nov 1;204:241-6. doi: 10.1016/j.jad.2016.06.040. Epub 2016 Jun 14. PMID 27450632
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2003-M-0211.html